CLINICAL TRIAL: NCT05442840
Title: Evaluation of Pharmacist Intervention and Education in a Patient-Centered, Multidisciplinary Approach for Individuals With Uncontrolled Type 2 Diabetes
Brief Title: Evaluation of Pharmacist Intervention for Individuals With Uncontrolled Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HS25460 (B2022:031)
Record Dates: First submitted 2022-06-20; First posted 2022-07-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 2 arms, either control or pharmacist intervention
Who Masked: Care Provider
Masking Description: The care provider (physician) will be aware the patient is participating in the study but will not be informed directly as to which arm they will be enrolled in, however if they review the electronic chart record they will be able to identify which arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): The participants in this arm will receive standard of care from their physician as they would have been doing previously. This still may involve blood work, referrals to other health providers (except pharmacist) and medication adjustments driven by the pharmacist.
- Pharmacist Intervention Arm (Active Comparator): The participants in this arm will receive standard of care from their physician in addition to pharmacist intervention. The pharmacist or pharmD intern leads the diabetes care for the patient typically, conducting a medication review, recommending medication changes, frequent follow up and requesting blood work and providing referrals to other health care providers as needed,which is standard care
  Interventions: Combination Product: Behavioral and drugs already approved and available for diabetes management

INTERVENTIONS:
Combination Product: Behavioral and drugs already approved and available for diabetes management — Pharmacists will review the patients information and medical history as well as drug coverage to discuss preferred treatment options to manage diabetes based on recommendations from Diabetes Canada treatment guidelines; all drugs have been approved and are available on the market; pharmacists will offer frequent follow up and provide basic diabetes education to the patient at each follow up appointment
  Arms: Pharmacist Intervention Arm

SUMMARY:
Type 2 diabetes is a chronic disease that can lead to a number of complications if uncontrolled and there is a projected increase of 33% patients living with diabetes over the next 10 years. There can be improvements to modifiable risk factors such as diet and exercise, in addition to medications. Treatment often involves a multidisciplinary approach with a physician, endocrinologist, dietitian, pharmacist and other support health professionals as required. This study will evaluate the effects of the pharmacists (or pharmD interns) intervention, looking at changes to the patients HbA1C, which is a measure of the patients blood glucose control over the previous 3 months as well as the patients understanding and comfort with managing their own diabetes via participant survey.

DETAILED DESCRIPTION:
Recruitment will begin in July 2022, potential participants can self-refer or another healthcare provider may discuss the study and provide contact information to the study team for all interested potential participants. These potential participants would then be screened for eligibility by the pharmacist or PharmD (Doctor of Pharmacy) Intern. The goal is to enroll 60 participants in the study. All participants must provide consent to participate and will be asked to complete a participant survey.

All participants who consented will then be randomized into a control group which will not receive pharmacist intervention during the study period, or the intervention group which will receive pharmacist/PharmD Intern led intervention which includes a medication review, optimizing medication treatment options and frequent follow up and diabetes education. The control group participants will be offered pharmacist intervention following the study period. All participants will be asked to complete a participant survey at the start and end of the study. All participants will also have standard care from their physicians and other healthcare team members as required which would be standard of practice. All participants would also be asked to repeat their blood work at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose primary care physician is within the Portage Clinic
* Adults (age 18 and older) with type 2 diabetes with HbA1C 10 % or above
* Patients whom have not had previous clinical pharmacist directed intervention
* Agree to participate in the study, including frequent follow up, blood glucose home monitoring as directed and repeat lab work
* Willing to consider medication adjustments as deemed appropriate
* Willing to review and sign the Research Participant Information and Informed Consent Form

Exclusion Criteria:

* Patients less than 18 years of age
* Patients with type 1 diabetes, pre-diabetes or gestational diabetes (or whom are pregnant)
* Patients whom have had recent or ongoing clinical pharmacist directed intervention or intensive health care professional monitoring and guidance
* Patients with HbA1C less than 10%
* Patients whom refuse medication adjustments
* Patients with severe renal impairment or receiving dialysis treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline Hemoglobin A1C (HbA1C) at 10 months | baseline and through study completion at 10 months approximately
  Measure of blood glucose control at the lab

SECONDARY OUTCOMES:
Participant Survey | baseline and through study completion at 10 months approximately
  Evaluating the patients knowledge of diabetes management, comfort with managing their own diabetes care, perception of the pharmacist's role
Modifiable Risk Factors -Cholesterol Level | baseline and through study completion at 10 months approximately
  evaluating changes in modifiable risk factors such as cholesterol levels reported in mmol/L
Modifiable Risk Factor - Body Mass Index | baseline and through study completion at 10 months approximately
  evaluating changes in modifiable risk factors such as weight and height which will be combined to report body mass index in kg/m^2
Modifiable Risk Factor - Blood Pressure | baseline and through study completion at 10 months approximately
  evaluating changes in modifiable risk factors such as blood pressure reported in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Portage Clinic, Portage la Prairie, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] APDS Diabetes Knowledge Questionnaire - Baker. (n.d.). Retrieved March 22, 2022, from https://www.baker.edu.au/-/media/documents/impact/ausdiab/questionnaires/ausdiab-diabetes-knowledge-questionnaire-2004.pdf?la=en
- [Background] Schmitt A, Gahr A, Hermanns N, Kulzer B, Huber J, Haak T. The Diabetes Self-Management Questionnaire (DSMQ): development and evaluation of an instrument to assess diabetes self-care activities associated with glycaemic control. Health Qual Life Outcomes. 2013 Aug 13;11:138. doi: 10.1186/1477-7525-11-138. PMID 23937988
- [Background] 36-Item Short form survey instrument (SF-36). RAND Corporation. (n.d.). Retrieved March 21, 2022, from https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/survey-instrument.html
- [Background] Jacobson, A. M., & Diabetes Control & Complications Trial Research Group. (1994). The Diabetes Quality of Life Measure. In C. Bradley (Ed.), Handbook of psychology and diabetes: A guide to psychological measurement in diabetes research and practice (pp. 65-87). Harwood Academic Publishers/Gordon.
- [Background] Bradley C: The Diabetes Treatment Satisfaction Questionnaire: DTSQ. In Handbook of Psychology and Diabetes: a guide to psychological measurement in diabetes research and practice. Edited by: Bradley C. Chur, Switzerland: Harwood Academic Publishers; 1994:111-132
- [Background] Syarifuddin S, Nasution A, Dalimunthe A, Khairunnisa. Impact of Pharmacist Intervention on Improving the Quality of Life of Patients with Type 2 Diabetes Mellitus. Open Access Maced J Med Sci. 2019 Apr 29;7(8):1401-1405. doi: 10.3889/oamjms.2019.140. eCollection 2019 Apr 30. PMID 31110593
- [Background] Bukhsh A, Nawaz MS, Ahmed HS, Khan TM. A randomized controlled study to evaluate the effect of pharmacist-led educational intervention on glycemic control, self-care activities and disease knowledge among type 2 diabetes patients: A consort compliant study protocol. Medicine (Baltimore). 2018 Mar;97(12):e9847. doi: 10.1097/MD.0000000000009847. PMID 29561461
- [Background] Abdulrhim S, Awaisu A, Ibrahim MIM, Diab MI, Hussain MAM, Al Raey H, Ismail MT, Sankaralingam S. Impact of pharmacist-involved collaborative care on diabetes management in a primary healthcare setting using real-world data. Int J Clin Pharm. 2022 Feb;44(1):153-162. doi: 10.1007/s11096-021-01327-x. Epub 2021 Oct 12. PMID 34637104
- [Background] Stading, J., Herrmann, J., Walters, R., Destache, C., Chock, A. (2009). Impact of Pharmacist Intervention on Diabetes Patients in an Ambulatory Setting. Diabetes Spectrum, Volume 22, Number 4, (241-246). https://diabetesjournals.org/spectrum/article/22/4/241/2441/Impact-of-Pharmacist-Intervention-on-Diabetes
- [Background] Jennings DL, Ragucci KR, Chumney EC, Wessell AM. Impact of clinical pharmacist intervention on diabetes related quality-of-life in an ambulatory care clinic. Pharm Pract (Granada). 2007 Oct;5(4):169-73. doi: 10.4321/s1886-36552007000400005. PMID 25170354
- [Background] Butt M, Mhd Ali A, Bakry MM, Mustafa N. Impact of a pharmacist led diabetes mellitus intervention on HbA1c, medication adherence and quality of life: A randomised controlled study. Saudi Pharm J. 2016 Jan;24(1):40-8. doi: 10.1016/j.jsps.2015.02.023. Epub 2015 Mar 6. PMID 26903767
- [Background] Shane-McWhorter L, McAdam-Marx C, Lenert L, Petersen M, Woolsey S, Coursey JM, Whittaker TC, Hyer C, LaMarche D, Carroll P, Chuy L. Pharmacist-provided diabetes management and education via a telemonitoring program. J Am Pharm Assoc (2003). 2015 Sep-Oct;55(5):516-26. doi: 10.1331/JAPhA.2015.14285. PMID 26359961
- See also: Diabetes Canada (2022, March). Diabetes in Manitoba: Backgrounder. Ottawa: Diabetes Canada; 2021. — https://www.diabetes.ca/DiabetesCanadaWebsite/media/Advocacy-and-Policy/Backgrounder/2021_Backgrounder_Manitoba_FINAL_1.pdf
- See also: Canadian Pharmacists Association, (2022, March). More and more Canadians say pharmacists play essential role in Canada's health care system, 2017. — https://www.pharmacists.ca/news-events/news/more-and-more-canadians-say-pharmacists-play-essential-role-in-canada-s-health-care-system/
- See also: The Canadian Diabetes Association. (2018). Diabetes Canada Clinical Practice Guidelines. Resources for People with Diabetes, Managing my Diabetes - My Action Plan. — https://guidelines.diabetes.ca/self-management/sme-action-plan
- See also: The Canadian Diabetes Association. (2015). Diabetes Canada Clinical Practice Guidelines. Patient resources, Medication sheet: SGLT2 Inhibitors — https://www.diabetes.ca/diabetescanadawebsite/media/managing-my-diabetes/tools%20and%20resources/medication-sheet-sglt2.pdf?ext=.pdf
- See also: The Canadian Diabetes Association. (2018). Diabetes Canada Clinical Practice Guidelines. Quick Reference Guide. — https://www.diabetes.ca/diabetescanadawebsite/media/health-care-providers/2018%20clinical%20practice%20guidelines/cpg-quick-reference-guide-web.pdf?ext=.pdf
- See also: The Canadian Diabetes Association. (2017). Tools and Resources, Insulin Prescription — https://www.diabetes.ca/DiabetesCanadaWebsite/media/Managing-My-Diabetes/Tools%20and%20Resources/insulin-prescription-fillable-EN.pdf?ext=.pdf
- See also: The Canadian Diabetes Association. (2018). Diabetes Canada Clinical Practice Guidelines. Tools and Resources, Insulin pen start checklist — https://www.diabetes.ca/DiabetesCanadaWebsite/media/Managing-My-Diabetes/Tools%20and%20Resources/insulin-pen-start-checklist.pdf?ext=.pdf
- See also: The Canadian Diabetes Association. (2018). Appendix 7: Therapeutic Considerations for Renal Impairment. (2018). Canadian Journal of Diabetes, 42 — https://www.diabetes.ca/DiabetesCanadaWebsite/media/Health-care-providers/2018%20Clinical%20Practice%20Guidelines/Appendix-7-therapeutic-considerations-for-renal-impairment.pdf?ext=.pdf
- See also: The Canadian Diabetes Association. (2020). 2020 Chapter Updates: Pharmacologic Glycemic Management of Type 2 Diabetes in Adults: 2020 Update — http://guidelines.diabetes.ca/cpg/chapter-13-2020-update
- See also: Health Canada. (April 2020). Side Effect Reporting Form — https://www.canada.ca/content/dam/hc-sc/migration/hc-sc/dhp-mps/alt_formats/pdf/medeff/report-declaration/ser-des_form-eng.pdf
- See also: The Canadian Diabetes Association. (2018). Appendix 6: Types of insulin. (2018). Canadian Journal of Diabetes, 42 — https://doi.org/10.1016/j.jcjd.2017.12.006